CLINICAL TRIAL: NCT04455750
Title: CASPAR - A Phase III Trial of Enzalutamide and Rucaparib as a Novel Therapy in First-Line Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Clinical Study Evaluating The Benefit of Adding Rucaparib to Enzalutamide for Men With Metastatic Prostate Cancer That Has Become Resistant To Testosterone-Deprivation Therapy
Acronym: CASPAR
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A031902; NCI-2020-02360 (Registry Identifier: NCI Clinical Trial Reporting Program); U10CA180821 (NIH)
Record Dates: First submitted 2020-06-17; First posted 2020-07-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Prostate Adenocarcinoma; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; Leuprolide; Goserelin; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (enzalutamide, rucaparib) (Experimental): Patients receive enzalutamide PO QD and rucaparib PO BID. Patients who did not undergo bilateral orchiectomy also receive ADT consisting of leuprolide acetate IM, goserelin acetate SC every 12 weeks or degarelix SC. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Enzalutamide; Drug: Rucaparib camsylate; Drug: Leuprolide Acetate; Drug: Goserelin Acetate; Drug: Degarelix; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (enzalutamide, placebo) (Active Comparator): Patients receive enzalutamide PO QD and placebo PO BID. Patients who did not undergo bilateral orchiectomy also receive ADT consisting of leuprolide acetate IM, goserelin acetate SC every 12 weeks or degarelix SC. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Enzalutamide; Drug: Placebo; Drug: Leuprolide Acetate; Drug: Goserelin Acetate; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Enzalutamide — Given PO
Drug: Rucaparib camsylate — Given PO
  Arms: Arm I (enzalutamide, rucaparib)
Drug: Placebo — Given PO
  Arms: Arm II (enzalutamide, placebo)
Drug: Leuprolide Acetate — Given IM
Drug: Goserelin Acetate — Given SC
Drug: Degarelix — Given SC
  Arms: Arm I (enzalutamide, rucaparib)
Other: Quality-of-Life Assessment — Ancillary studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized, placebo-controlled phase III trial is evaluating the benefit of rucaparib and enzalutamide combination therapy versus enzalutamide alone for the treatment of men with prostate cancer that has spread to other places in the body (metastatic) and has become resistant to testosterone-deprivation therapy (castration-resistant). Enzalutamide helps fight prostate cancer by blocking the use of testosterone by the tumor cells for growth. Poly adenosine diphosphate (ADP)-ribose polymerase (PARP) inhibitors, such as rucaparib, fight prostate cancer by prevent tumor cells from repairing their DNA. Giving enzalutamide and rucaparib may make patients live longer or prevent their cancer from growing or spreading for a longer time, or both. It may also help doctors learn if a mutation in any of the homologous recombination DNA repair genes is helpful to decide which treatment is best for the patient.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare radiographic progression-free survival (rPFS) and overall survival (OS) with enzalutamide and rucaparib camsylate (rucaparib) versus enzalutamide alone for patients with metastatic castration resistant prostate cancer commencing first-line therapy.

II. (PK substudy) To evaluate the safety and tolerability of rucaparib and enzalutamide combination III. (Quality of life substudy) To compare quality of life as measured by FACT-P Trial Outcome Index in patients with mCRPC who receive enzalutamide plus rucaparib vs enzalutamide alone at the 12-month time point (primary QOL timepoint).

SECONDARY OBJECTIVES:

I. To compare rPFS and OS with enzalutamide and rucaparib versus enzalutamide alone within homologous-recombination repair (HRR) aberrant and wild-type patients.

II. To evaluate the effects of concurrent administration of rucaparib on time to unequivocal clinical progression.

III. To evaluate the effects of concurrent administration of rucaparib on best radiographic response using Prostate Cancer Working Group 3 (PCWG3) criteria.

IV. To evaluate the effects of concurrent administration of rucaparib on duration of overall response.

V. To evaluate the effects of concurrent administration of rucaparib on prostate specific antigen (PSA) response rate.

VI. To evaluate the effects of concurrent administration of rucaparib on best response by serum PSA by months 7 and 13.

VII. To evaluate the effects of concurrent administration of rucaparib on time to first symptomatic skeletal event (SSE).

VIII. To evaluate the effects of concurrent administration of rucaparib on safety and tolerability as measured by National Cancer Institute (NCI) Common Toxicity Criteria; and trial discontinuation for treatment emergent toxicities.

IX. To compare performance of plasma-based and tissue-based genomic profiling in detection of homologous-recombination repair mutation (HRRm) in metastatic castration-resistant prostate cancer (mCRPC).

OUTLINE:

In the randomized, placebo-controlled phase III study, patients will be randomized to 1 of 2 arms:

ARM I: Patients will receive enzalutamide orally (PO) once daily (QD) and rucaparib PO twice daily (BID). Patients who did not undergo bilateral orchiectomy will also receive androgen deprivation therapy (ADT) consisting of leuprolide acetate intramuscularly (IM), goserelin acetate subcutaneously (SC) every 12 weeks or degarelix SC. Cycles will repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients will receive enzalutamide PO QD and placebo PO BID. Patients who did not undergo bilateral orchiectomy will also receive ADT consisting of leuprolide acetate IM, goserelin acetate SC every 12 weeks or degarelix SC. Cycles will repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After the completion of study treatment, patients will be followed every 3 months for 2 years, then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic/cytologic documentation of prostate adenocarcinoma
* Adequate archival tumor specimen or archival slides must be available to be tested as part of the trial screening (most recent metastatic site biopsy preferred, but primary prostate biopsy allowed if metastatic biopsy is not available or inadequate. A new biopsy is not required for pre-registration in the trial as long as sufficient archival tissue is available). Due to significant variability between tests, results from an existing targeted next-generation exome sequencing test may not be used for this trial
* Progressive disease must be demonstrated at study entry while the patient is on continuous androgen deprivation therapy (ADT) or status post orchiectomy. Progressive disease is defined as one or more of the following criteria:

  * PSA progression, defined by at least 2 consecutive rising PSA values at a minimum of 1-week intervals with the most recent PSA value being 1.0 ng/mL or higher, if confirmed PSA rise is the only indication of progression. Patients who received an anti-androgen must have PSA progression after withdrawal of anti-androgen therapy (>=4 weeks since last flutamide, bicalutamide or nilutamide, apalutamide or darolutamide)
  * Radiographic progression per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 for soft tissue lesions
  * Bone metastasis progression per Prostate Cancer Working Group 3 (PCWG3) criteria
* Measurable or non-measurable metastatic disease
* No prior therapy for metastatic castration-resistant prostate cancer, defined as a treatment given for prostate cancer with radiographically-detectable metastasis and a serum testosterone level less than 50 ng/dl (1.73 nmol/L) at the time of registration
* >= 2 weeks or 5 half-lives (whichever is shorter) since prior therapy with flutamide, dutasteride, bicalutamide, niltamide, finasteride, aminoglutethimide, estrogens, cytoproterone, chemotherapy, abiraterone, apalutamide, or darolutamide
* >= 4 weeks or 5 half-lives (whichever is shorter) since any prior investigational therapy
* >= 4 weeks since a major surgery or radiation
* No prior therapy with enzalutamide, rucaparib or any other PARP inhibitor, or platinum chemotherapy
* Prior docetaxel and/or novel anti-androgen use is allowed only if given in the hormone-sensitive non-metastatic or metastatic, or castration-resistant non-metastatic disease setting
* Patient must have discontinued all previous treatments for cancer (except ADT and bone anti-responsive therapies such as denosumab or zoledronic acid) and must have recovered from all acute side effects of prior therapy or surgical procedures to =< grade 1 or baseline prior to randomization, with the exception of fatigue, alopecia or peripheral neuropathy
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 10 g/dL
* Serum testosterone =< 50 ng/dl (=< 1.73 nmol/L)
* Serum creatinine =< 1.5 x upper limit of normal (ULN)
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate transaminase (AST)/alanine transferase (ALT) =< 2.5 x upper limit of normal (ULN)
* No clinically suspected central nervous system (CNS) (leptomeningeal or parenchymal) metastases. Patients with a history of CNS metastasis(s) will be allowed as long (1) as the metastatic site(s) were adequately treated as demonstrated by clinical and radiographic improvement, AND (2) the patient has recovered from the intervention (no residual adverse events > Common Terminology Criteria for Adverse Events [CTCAE] grade 1), AND (3) the patient has remained without occurrence of new or worsening CNS symptoms for a period of 28 days prior to pre-registration
* No known or suspected history of cytopenia (low white blood cell [WBC], hemoglobin or platelet count) of greater than 3 months duration with an unknown cause, myelodysplastic syndrome, or hematologic malignancies
* No blood product transfusion, granulocyte/granulocyte-macrophage-colony stimulating factor (G-CSF/GM-CSF), or erythropoietin/thrombopoietin use within 14 days of pre-registration
* No history of syncope of cardiovascular etiology, uncontrolled cardiac arrhythmia, history of Mobitz II second degree or third degree heart block without a permanent pacemaker in place, myocardial ischemia or infarction, severe or unstable angina, New York Heart Association (NYHA) class II to IV heart failure, or stroke/transient ischemic attack (TIA) within the past 3 months
* No history of seizure or any condition that may increase the patient's seizure risk (e.g., prior cortical stroke, significant brain trauma) within 2 years
* No clinically active or chronic liver disease resulting in moderate/severe hepatic impairment (Child-Pugh class B or C), ascites, coagulopathy or bleeding due to liver dysfunction
* No clinical, laboratory or radiographic evidence of an active bacterial, fungal, or viral infection requiring treatment at the time of registration
* No planned palliative procedures for alleviation of bone pain such as radiation therapy or surgery
* No untreated spinal cord compression or evidence of spinal metastases with a risk of impending fracture or spinal cord compression
* No known or suspected contraindications or hypersensitivity to enzalutamide, rucaparib, or to any of the excipients
* No known or suspected gastrointestinal disorder affecting absorption of oral medications
* No prior malignancy for which the last treatment was given within the past 2 years, or any active concurrent malignancy with the exception of non-melanomatous localized skin cancers (such as squamous or basal cell carcinoma of the skin)
* Any concomitant medications that are strong inhibitors of CYP2C8 or inducers of CYP3A4 cytochrome enzymes must be discontinued prior to registration. Dose adjustments per Food and Drug Administration (FDA) label or clinical judgement should be considered for any concomitant medications that are moderate inhibitors of CYP2C8 or inducers of CYP3A4 cytochrome enzymes
* Any concomitant medications that are substrates of CYP3A4, CYP2C9 and CYP2C19 cytochrome enzymes should be monitored closely per clinical judgement of the treating physician

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Radiographic progression-free survival (rPFS) | Up to 5 years post treatment
  Radiographic progression-free survival (rPFS) is defined as the time from randomization to date of disease progression or death due to any cause. rPFS time will be compared between the treatment arms using a log-rank test. Median times per treatment arms will be reported.
Overall survival (OS) | Up to 5 years post treatment
  Overall survival is defined as the time from randomization to death due to any cause. Overall survival time will be compared between the treatment arms using a log-rank test. Median times per treatment arms will be reported.

SECONDARY OUTCOMES:
Radiographic progression-free survival (rPFS) within HRRm status | Up to 5 years post treatment
  Defined as the time from randomization to date of disease progression or death due to any cause. rPFS time will be compared between the treatment arms using a log-rank test. Median times per treatment arms will be reported.
Time to unequivocal clinical progression | Up to 5 years post treatment
  Defined as deterioration in clinical status clearly attributable to prostate cancer progression with occurrence of cancer pain requiring initiation of chronic administration of opiate analgesia, or an immediate need to re-initiate cytotoxic chemotherapy, radiation therapy or surgical intervention for disease-progression related events; or deterioration of Eastern Cooperative Oncology Group (ECOG) performance status to 3 or greater. Time to unequivocal clinical progression will be compared between the treatment arms using a log-rank test. Median times per treatment arms will be reported.
Overall survival by HRRm status | Up to 5 years post treatment
  Defined as the time from randomization to death due to any cause.Overall survival time will be compared between the treatment arms using a stratified (by HRRm status) log-rank test. Median times per treatment arms/HRRm status will be reported.
Overall response rate | Up to 1 year after completion of treatment
  Defined as confirmed radiographic complete response or partial response. The proportion of patients with confirmed radiographic response or partial response will be compared between the treatment arms with a chi-square test (or Fisher's exact test if more appropriate).
Duration of overall response | Up to 1 year after completion of treatment
  Defined as the time from documentation of a radiographic response to disease progression. Duration of response time will be compared between the treatment arms using a log-rank test. Median times per treatment arms will be reported.
Prostate specific antigen (PSA) response rate | Up to 1 year after completion of treatment
  Defined as >= 50% reduction in PSA from baseline. The proportion of patients with PSA response will be compared between the treatment arms with a chi-square test (or Fisher's exact test if more appropriate).
Best response by serum prostate specific antigen (PSA) | At 7 and 13 months from the start of treatment
  Defined as best percentage PSA decline from baseline to 7 and 13 months. The percent PSA decline will be compared between treatment arms with a Wilcoxon rank sum test.
Time to first symptomatic skeletal event (SSE) | Up to 5 years after completion of treatment
  Defined as the time to first use of external-beam radiation therapy to relieve skeletal symptoms, new symptomatic pathologic vertebral or nonvertebral bone fractures, spinal cord compression, or tumor-related orthopedic surgical intervention. Time to first SSE will be compared between the treatment arms using a log-rank test. Median times per treatment arms will be reported.
Incidence of adverse events | Up to 1 year after completion of treatment
  Frequency as measured by National Cancer Institute (NCI) Common Toxicity Criteria. The proportion of patients experiencing at least one grade 3+ adverse event will be compared between the treatment arms with a chi-square test (or Fisher's exact test if more appropriate).
Discontinuation for treatment emergent toxicities | Up to 1 year after completion of treatment
  The proportion of patients who discontinued treatment for emergent toxicities will be compared between the treatment arms with a chi-square test (or Fisher's exact test if more appropriate).

OTHER OUTCOMES:
Quality of life | 12 months
  Measured by change from baseline to 12 months of the Trial Outcome Index of the Functional Assessment of Cancer Therapy-Prostate (FACT-P) patient-reported outcome questionnaire.
Quality of life | 12 months
  Measured by change from baseline to 12 months of the Utility Score of the European Quality of Life Five Dimension Five Level (EQ-5D-5L) patient-reported outcome questionnaire.
Laboratory correlative science | Up to 1 year after completion of treatment
  Area under curve for plasma-based and tissue-based genomic profiling in detection of HRRm in mCRPC.
Laboratory correlative science | Up to 1 year after completion of treatment
  The proportion of patients with homologous-recombination repair (HRR) alterations at baseline who develop HRR reversion/function restoring alterations after initiation of treatment in each arm with a chi-square test (or Fisher's exact test if more appropriate).

CONTACTS AND LOCATIONS:
Overall Officials: Arpit Rao, MD, Study Chair — Baylor College of Medicine
Locations (414):
- United States (414):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Sharp Memorial Hospital, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Northbay Cancer Center, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Augusta Oncology Associates PC-D'Antignac, Augusta, Georgia
  - Augusta Oncology Associates PC-Wheeler, Augusta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola Medicine Homer Glen, Homer Glen, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ascension Borgess Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - The New York Hospital Medical Center of Queens, Flushing, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Queens Hospital Center, Jamaica, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Nyack Hospital, Nyack, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Wake Forest Baptist Health - Wilkes Medical Center, Wilkesboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Southpointe-Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Avera Cancer Institute at Yankton, Yankton, South Dakota
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Centra Lynchburg Hematology-Oncology Clinic Inc, Lynchburg, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - FHCC Overlake, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Seattle Cancer Care Alliance at EvergreenHealth, Kirkland, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - FHCC at Northwest Hospital, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: Yes